CLINICAL TRIAL: NCT04508686
Title: Phase 1 Trail to Observe Safety and Efficacy of Metronomic Capecitabine Plus PD-L1 Antibody Camrelizumab as Third-line Regimen to Treat HER2 Negative Advanced Gastric Cancer Patients
Brief Title: Combination of Metronomic Capecitabine With Camrelizumab for Treatment of Refractory Solid Tumor Trial (Cohort 1)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Jun Zhang, Chair of Department of Oncology, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: McCrest
Record Dates: First submitted 2020-08-06; First posted 2020-08-11 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Advanced Cervical Cancer
MeSH Terms: interventions — Capecitabine; camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Capecitabine 500mg bid. po. Camrelizumab 200mg ivgtt. d1 q2w
  Interventions: Drug: Capecitabine, camrelizumab

INTERVENTIONS:
Drug: Capecitabine, camrelizumab — This is a single-arm study with all patients receiving these two drugs.

SUMMARY:
This is a single center phase 1 trail to observe safety and efficacy of metronomic capecitabine plus PD-L1 antibody camrelizumab as third-line regimen to treat HER2 negative advanced gastric cancer patients.

This study is one of the cohorts of a multi-cohort trial called Combination of Metronomic capecitabine with Camrelizumab for treatment of refractory solid tumor (McCrest) trial.

DETAILED DESCRIPTION:
HER2 negative advanced gastric cancer patients who have disease progression after two standard regimens will be treated by metronomic capecitabine plus camrelizumab. Metronomic capecitabine will be given as fixed dose (500mg bid) orally. Camrelizumab will be given two-weekly (200mg once) intravenously. This regimen will be administered until progression of disease, intolerable toxicity or withdraw of consent.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female patients aged≥18 years.
2. Histologically confirmed gastric or gastric esophageal junction adenocarcinoma, without uncontrolled pleural effusion or ascites.
3. Patients with advanced or metastatic disease who have disease progression after two standard regimens, with measurable or unmeasurable lesions.
4. HER2 negative, MSS or pMMR.
5. ECOG performance status 0 or 2, expected lifetime≥3 months.
6. Adequate organ function: Absolute neutrophil count (ANC) ≥1.5x109/L, White blood count ≥3.5x109/L, Platelets ≥75x109/L, Hemoglobin (Hb) ≥70g/L, ALT/AST ≤2.5x ULN (for patient with liver metastasis ALT/AST ≤5x ULN), Serum bilirubin ≤1.5x ULN, Serum creatinine ≤1.5x ULN.
7. HBV infected patients (inactive/asymptomatic carrier, chronic or active) with HBV DNA<500IU/ml (or 2500 copies/ml).
8. Pregnancy test of female patients with fertile activity should be negative within 7 days before enrollment. Patients should keep contraception during treatment.
9. Willingness and ability to comply with the protocol for the duration of the study including scheduled visits, examinations, investigations and treatment plans with informed consent form.

Exclusion Criteria:

1. Pregnancy or children bearing potential.
2. brain or meningeal metastasis.
3. With second primary malignant diseases.
4. With uncontrolled auto-immune diseases, interstitial pneumonia, ulcerative colitis, or patients who should receive long-term glucocorticoid treatment (>10mg/d prednisone).
5. With uncontrollable complications
6. Inadequate organ function
7. Conditions which impact on pill taking (dysphagia, chronic diarrhea, bowel obstruction).
8. known hypersensitivity reaction to any of the study drugs or components.
9. Other unsuitable conditions determined by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Safety: adverse events as assessed by CTCAE v5.0 | 48 months

SECONDARY OUTCOMES:
Progression free survival | 48 months
Overall survival | 48 months
Objective response rate | 48 months
Disease control rate | 48 months
Duration of response | 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, MD & Ph. D, Principal Investigator — Ruijin Hospital
Locations (1):
- Department of Oncology, Ruijin Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou C, Yin Y, Shangguan C, Wu Q, Cai Q, Xi W, Guo L, Jiang J, Shi M, Wu J, Ji J, Zhang X, Sun Y, Rensen SSM, Damink SWMO, Zhu Z, Zeng R, Zhang J. Lipid metabolism associated with efficacy of metronomic capecitabine and camrelizumab in gastrointestinal cancer: an exploratory clinical trial. BMC Med. 2025 Oct 21;23(1):572. doi: 10.1186/s12916-025-04377-4. PMID 41121239